CLINICAL TRIAL: NCT05348213
Title: Clinical Study of Efficacy and Safety of Novel Targeted Drugs Combined With R-ICE Regimen in the Treatment of Relapsed and Refractory Diffuse Large B-cell Lymphoma
Brief Title: Novel Targeted Drugs Combined With R-ICE Regimen in Relapsed and Refractory Diffuse Large B-cell Lymphoma
Acronym: R-ICE+X
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-ICE+X
Record Dates: First submitted 2022-01-10; First posted 2022-04-27 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B Cell Lymphoma; R-ICE+X
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; Decitabine; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; tofacitinib; pomalidomide; protease resembling ICE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-ICE+X (Experimental): R-ICE plus novel targeted drugs
  Interventions: Drug: Zanubrutinib plus R-ICE; Drug: Decitabine plus R-ICE; Drug: Chidamide plus R-ICE; Drug: Tofacitinib plus R-ICE; Drug: Pomalidomide plus R-ICE

INTERVENTIONS:
Drug: Zanubrutinib plus R-ICE — Zanubrutinib 160mg/bid PO D1-21 Rituximab 375mg/m2 IV D0 Ifosfamide 1500mg/m2 IV D1-3 Carboplatin AUC×[GFR(ml/min) + 25] mg/d,AUC=5 IV D2 Etoposide 100 mg/m2 IV D1-3
  Other Names: ZR-ICE
Drug: Decitabine plus R-ICE — Decitabine 10mg/m2 IV D1-5 Rituximab 375mg/m2 IV D0 Ifosfamide 1500mg/m2 IV D1-3 Carboplatin AUC×[GFR(ml/min) + 25] mg/d,AUC=5 IV D2 Etoposide 100 mg/m2 IV D1-3
  Other Names: DR-ICE
Drug: Chidamide plus R-ICE — Chidamide 20mg/d PO D1、4、8、11 Rituximab 375mg/m2 IV D0 Ifosfamide 1500mg/m2 IV D1-3 Carboplatin AUC×[GFR(ml/min) + 25] mg/d,AUC=5 IV D2 Etoposide 100 mg/m2 IV D1-3
  Other Names: CR-ICE
Drug: Tofacitinib plus R-ICE — Tofacitinib 5mg/bid PO D1-10 Rituximab 375mg/m2 IV D0 Ifosfamide 1500mg/m2 IV D1-3 Carboplatin AUC×[GFR(ml/min) + 25] mg/d,AUC=5 IV D2 Etoposide 100 mg/m2 IV D1-3
  Other Names: TR-ICR
Drug: Pomalidomide plus R-ICE — Pomalidomide 4mg/d PO D1-10 Rituximab 375mg/m2 IV D0 Ifosfamide 1500mg/m2 IV D1-3 Carboplatin AUC×[GFR(ml/min) + 25] mg/d,AUC=5 IV D2 Etoposide 100 mg/m2 IV D1-3
  Other Names: PR-ICE

SUMMARY:
A single-center, open, single-arm clinical study of the efficacy and safety of a novel targeted agent in combination with R-ICE in the treatment of relapsed and refractory diffuse Large B-cell lymphoma.

DETAILED DESCRIPTION:
Refractory recurrence of patients with diffuse large B cell lymphoma inclusion/exclusion standard subjects in a signed written informed consent, according to the results of genotyping, divided the patients into MCD, TP53, BN2, EZB, ST2, NOS, N1, a total of 7 kinds of types. New targeted drugs were added based on typing results: Zanubrutinib for MCD and BN2, Decitabine for TP53, Chidamide for EZB, Tofacitinib for ST2, and Pomalidomide for N1 and NOS. After 3 courses of treatment, PET-CT was used to evaluate the efficacy. Patients with CR/PR, aged ≤65 years, qualified and willing for transplantation, were treated with autologous hematopoietic stem cell transplantation (ASCT); Patients who did not meet the above requirements or failed to collect autologous hematopoietic stem cells were placed on new targeted drug maintenance therapy for up to 12 months; If patients were evaluated as SD and PD after 3 cycles, they were treated with other regiments. New targeted drugs combined with R-ICE and ASCT were evaluated every 3 months in the first year and every 6 months in the second and third years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* DLBCL was confirmed by histology according to world Health Organization (WHO) disease classification (excluding primary central lymphoma and HIV-associated lymphoma);
* There are evaluable lesions detected by PET/CT;
* Life expectancy of more than 3 months;
* Prior treatment with sufficient first-line anti-lymphoma therapy, no remission within 90 days of the last administration, or disease progression after sufficient first-line anti-lymphoma therapy, and no current anti-lymphoma therapy (≥2 weeks since the last anti-lymphoma therapy). Patients were allowed to receive hormone drugs or rituximab at least 1 week after enrollment for symptom control reasons;
* 18≤ age ≤75 years old, male and female;
* ECOG 0-2 points;
* No serious organic lesions in the main organs, meeting the requirements of the following laboratory examination indicators (conducted within 7 days before treatment) :

  ① Absolute value of neutrophil count ≥1500/mm3; Platelet count ≥75,000/mm3

  ② Total bilirubin ≤2× upper limit of normal value (ULN)

  ③ Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (serum glutamate pyruvate aminotransferase [SGPT]) ≤3× upper limit of normal value (ULN)

  ④ the creatinine clearance rate was ≥60ml/min

  ⑤ No cardiac dysfunction
* If the subject is of reproductive age and requires effective contraception, he/she agrees to comply with all contraceptive requirements: 1) there are fertile women have to decide, at the same time take two reliable contraceptive methods (a kind of high efficient contraceptives - tubal ligation, intrauterine contraceptive device, hormone (birth control pills, needle, patch, vaginal ring or implants) or partner vasectomy, another effective birth control method -- men or synthetic rubber condom, diaphragm or cervical cap). 2) Unless hysterectomy, effective contraception is required even if there is a history of infertility;
* Fertile men must always use rubber or synthetic condoms when having sexual contact with fertile women during the use of this product and within 28 days of discontinuation of this product, even if they have successfully vasectomy; The subjects knew the characteristics of the disease, voluntarily joined the study, received treatment and follow-up, and the informed consent was signed by the subjects themselves or their guardians and impartial witnesses.

Exclusion Criteria:

* Pregnant or lactating women (lactating women must agree not to breastfeed while taking pomadomide);
* Known hepatitis B (HBV), hepatitis C (HCV) infection (HBV infection refers to HBV-DNA > detectable limit); And other acquired, congenital immune deficiency disorders, including but not limited to HIV-infected persons;
* Subjects with a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 12 months;
* Bone marrow failure, defined as ANC<1500/mm3 or platelet <75,000/mm3, unless hematologic changes are thought to be associated with lymphomas infiltrating the bone marrow;
* Clinically significant heart disease, including unstable angina, acute myocardial infarction 6 months before enrollment, congestive heart failure (NYHA) heart function grade III or IV; Or left ventricular ejection fraction <50%;
* Lymphoma with central nervous system (CNS) involvement;
* Those who are known to be allergic to the test drug ingredients;
* Those who have received grade II or above surgery within three weeks before treatment;
* Patients who have received organ transplants;
* Has been diagnosed with or is being treated for malignancy other than lymphoma, except for:

  ① They have received therapeutic treatment and have not had known active disease malignancy for ≥5 years prior to enrollment;

  ② Basal cell carcinoma of the skin (except melanoma) without signs of disease after adequate treatment;

  ③ Cervical carcinoma in situ without signs of disease after adequate treatment.
* With severe infection;
* Substance abuse, medical, psychological, or social conditions that may interfere with the subjects' participation in the study or evaluation of the study results; The researchers deemed unsuitable for the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate after 3 cycle chemotherapy | At the end of cycle 3 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Objective remission rate after 3 cycle chemotherapy | At the end of cycle 3 (each cycle is 21 days)
  Percentage of participants with complete response or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
2 year progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
2 year overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.
Chemotherapy-related adverse reactions | At the end of cycle 3 (each cycle is 21 days)
  Any harmful reaction that occurs during the treatment of a disease according to the normal usage and dosage of a drug, which is unrelated to the purpose of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No